CLINICAL TRIAL: NCT01908257
Title: A Phase 1, Open-Label, Drug-Drug Interaction Study to Evaluate the Potential Effects of Ranitidine on the Pharmacokinetics of Lesinurad in Healthy Adult Male Subjects
Brief Title: Lesinurad Interaction Study With Ranitidine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RDEA594-127
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Healthy
MeSH Terms: interventions — lesinurad; Ranitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 fasted (Experimental): Day 1: Lesinurad 400 mg once daily (qd)
  Day 5: Ranitidine 150 mg twice daily (bid)
  Day 6: Lesinurad 400 mg (qd) + ranitidine 150 mg (bid). Ranitidine dosed at -2 hours predose and 12 hours postdose of lesinurad.
  Day 7: Ranitidine 150 mg (bid)
  Interventions: Drug: lesinurad 400 mg; Drug: ranitidine 150 mg; Drug: lesinurad 400 mg + ranitidine 150 mg
- Sequence 2 fasted (Experimental): Day 1: Ranitidine 150 mg (bid)
  Day 2: Lesinurad 400 mg (qd) + ranitidine 150 mg (bid). Ranitidine dosed at -2 hours predose and 12 hours postdose of lesinurad
  Day 3: Ranitidine 150 mg (bid)
  Day 7: Lesinurad 400 mg (qd)
  Interventions: Drug: lesinurad 400 mg; Drug: ranitidine 150 mg; Drug: lesinurad 400 mg + ranitidine 150 mg

INTERVENTIONS:
Drug: lesinurad 400 mg
Drug: ranitidine 150 mg
Drug: lesinurad 400 mg + ranitidine 150 mg

SUMMARY:
This is a drug-drug interaction study in healthy volunteers to evaluate the potential pharmacokinetic (PK) effects of ranitidine on lesinurad.

DETAILED DESCRIPTION:
This study will evaluate the potential effect of ranitidine on the pharmacokinetics of lesinurad. An earlier study demonstrated an effect on lesinurad PK in the presence of both calcium-containing and magnesium- and aluminum-containing antacids. The current study will assess whether raising gastric pH, without the presence of these cations, affects lesinurad PK and PD under the fasted state. If an impact is seen, then the optional second cohort will be conducted under the fed state.

ELIGIBILITY:
Inclusion Criteria:

* body weight ≥ 50 kg (110 lbs) and body mass index ≥ 18 and ≤ 30 kg/m2.
* Screening sUA value ≤ 7.0 mg/dL.
* free of any clinically significant disease that requires a physician's care and/or would interfere with study evaluations or procedures.
* Subject has no clinically relevant abnormalties in vital signs, ECG, physical examination or safety laboratory values per the Investigator's judgment.

Exclusion Criteria:

* history or clinical manifestations of significant metabolic, hematological, pulmonary, cardiovascular, gastrointestinal, neurologic, hepatic renal,urological, or psychiatric disorders.
* history or suspicion of kidney stones.
* undergone major surgery within 3 months prior to Day 1.
* donated blood or experienced significant blood loss (> 450 mL) within 12 weeks prior to Day 1 or gave a plasma donation within 4 weeks prior to the Screening visit.
* inadequate venous access or unsuitable veins for repeated venipuncture.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
PK profile of lesinurad from plasma and urine | Days 1 and 6 (Sequence 1) or Days 2 and 7 (Sequence 2)
  Profile in terms of Cmax, Tmax, AUC, CL/F, t1/2
  Cmax: maximum concentration; Tmax: time to reach max plasma concentration; AUC: area under the concentration-time curve; CL/F: total body clearance corrected for bioavailability; t1/2: apparent terminal half-life

SECONDARY OUTCOMES:
Incidence of Adverse Events and Changes in Laboratory, Electrocardiogram, and Vital Signs Parameters | 6 weeks
PD profile of lesinurad from serum | Days 1 and 6 (Sequence 1) or Days 2 and 7 (Sequence 2)
  Profile in terms of serum urate concentration

CONTACTS AND LOCATIONS:
Overall Officials: S. Bradley, MD, Study Director — Ardea Biosciences, Inc.
Locations (1):
- Cypress, California, United States